CLINICAL TRIAL: NCT07379164
Title: Psychophysiological Restorative Effects of Green Exercise: A Randomized Controlled Trial
Brief Title: Psychophysiological Effects of Green Exercise in Outdoor Green vs. Indoor Control
Acronym: GREEN-OI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lincoln University College (Other)
Collaborators: Wuhan Technical University (Unknown)
Responsible Party: Principal Investigator, Linjun Liu, Doctoral Researcher, Lincoln University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WTU-IRB-2025-0113
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Psychological Stress; Mental Fatigue; Cognitive Dysfunction; Emotional Well-being; Healthy Volunteers
Keywords: Green Exercise; Nature-based Interventio; Attention Restoration Theory; Psychophysiological Restoration; Urban Health
MeSH Terms: conditions — Stress, Psychological; Mental Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized, two-arm, parallel-group controlled trial. Participants are randomly assigned to either the Outdoor Green group or the Indoor Control group with a 1:1 allocation ratio. Each participant stays in their assigned group throughout the study duration and completes a standardized 30-minute walking task in their respective environment (an outdoor forest park versus an indoor laboratory).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor Green Group (Experimental): Participants in this arm perform a standardized 30-minute walk at a moderate pace along a pre-defined route in an outdoor green enviroment. This arm focuses on the effects of exposure to natural environmental stimuli.
  Interventions: Behavioral: Outdoor Green Group
- Indoor Control Group (Active Comparator): Participants walk on a treadmill at a fixed moderate speed (4.0-5.5 km/h) with a 1% incline. This specific incline is used to compensate for the lack of air resistance indoors and to more accurately match the physiological energy expenditure of outdoor ground walking.
  Interventions: Behavioral: Indoor Control Group

INTERVENTIONS:
Behavioral: Outdoor Green Group — Participants perform a supervised 30-minute walk at a moderate pace (4.0-5.5 km/h) along a pre-defined 2.5 km loop trail within a suburban forest park. The environment is characterized by high canopy cover (>60%) and diverse natural vegetation. To ensure consistency, all sessions are conducted under stable weather conditions (Temperature: 20-26°C; Humidity: 40-60%). Participants walk individually to prevent social interaction, ensuring the restorative experience is derived solely from the individual-nature interaction.
  Arms: Outdoor Green Group
Behavioral: Indoor Control Group — Participants perform a 30-minute walk on a treadmill in a windowless indoor laboratory. To ensure consistency with the outdoor environment, the laboratory is climate-controlled with a temperature range of 20-26°C and humidity of 40-60%. The treadmill is set to a fixed moderate speed (4.0-5.5 km/h) with a 1% incline. The 1% incline is specifically applied to compensate for the lack of air resistance indoors and to accurately match the physiological energy expenditure and biomechanical demands of outdoor ground walking. The laboratory walls are neutral-colored to eliminate visual nature stimuli.
  Arms: Indoor Control Group

SUMMARY:
Core Purpose: Researchers want to learn if walking in an outdoor green environment helps people recover from mental tiredness and stress better than walking indoors. This study investigates how a 30-minute walk in an outdoor green setting affects the mind and body compared to a 30-minute walk on a treadmill in a room without windows.

The Study Process: The study included 80 healthy young adults between the ages of 18 and 35. Researchers randomly split the participants into two groups.

1. The Outdoor Green group: Participants walked for 30 minutes on a path in an outdoor green environment.
2. The Indoor Control group: This group walked for 30 minutes on a treadmill in a windowless room.

What is Being Measured: To understand how the environment helps the brain recover, researchers used a "Sensory-to-Appraisal" model to measure several factors.

1. Information Harvesting: Researchers used a new tool called the Nature Sensory Sensitivity Index (NSSI). This measures how well participants notice and "capture" sensory details from their surroundings, like the sounds of birds or the textures of plants.
2. Restorative Feelings: Using the Perceived Restorativeness Scale (PRS), participants reported if they felt the environment helped them "get away" from daily stress and if the setting was interesting or beautiful.
3. Overall Mood Changes (POMS TMD): Researchers used the Profile of Mood States (POMS) to calculate a Total Mood Disturbance (TMD) score. This helps show if participants feel less tense, angry, or tired, and more energetic after the walk.
4. Connection to Nature (NR): Researchers measured each participant's Nature Relatedness (NR). This describes how much a person naturally feels connected to the natural world, which may influence how much they benefit from the green walk.
5. Attention and Thinking: Participants performed a "Digit Span Task" (repeating sequences of numbers) to test if their focus improved.
6. Physical Stress: The study used objective markers, including salivary cortisol (a stress hormone) and heart rate variability (a measure of how the nervous system relaxes).

Why This Matters: The goal of this research is to see if actively noticing an outdoor green environment (sensory harvesting) is the "key" that unlocks mental recovery. By comparing the Outdoor Green group with the Indoor Control group, this study helps us understand why nature is good for public health and how to design better spaces for stress relief.

DETAILED DESCRIPTION:
Study Overview and Theoretical Framework This randomized controlled trial (RCT) aims to investigate the psychophysiological restorative effects of green exercise. The study is grounded in Attention Restoration Theory (ART) and Stress Recovery Theory (SRT). It specifically tests a "Sensory-to-Appraisal" model, which proposes that the restorative benefits of nature are driven by an initial stage of objective sensory information harvesting, followed by subjective restorative appraisal.

Experimental Design A total of 80 healthy young adults (aged 18-35) were recruited and randomly assigned to one of two groups with a 1:1 allocation ratio.

1. The Outdoor Green group: Participants performed a standardized 30-minute walk along a pre-defined route in a forest park environment.
2. The Indoor Control group: Participants performed a 30-minute walk on a treadmill in a controlled laboratory setting (windowless room, neutral environment) at a self-selected moderate pace to match the physical intensity of the outdoor group.

Experimental Procedure The experiment followed a five-stage longitudinal design.

1. Baseline (T0): Collection of demographic data, Nature Relatedness (NR) scales, and initial physiological/psychological measurements.
2. Stress Induction: Participants underwent a cognitive stressor to induce mental fatigue and psychological stress.
3. Intervention (T1): The 30-minute walking intervention in the assigned environment.
4. Post-Intervention (T2): Immediate post-test measurements including sensory harvesting (NSSI), perceived restorativeness (PRS), and emotional states.
5. Recovery Monitoring: Follow-up assessment of cognitive function and physiological recovery markers.

Key Measures

1. Sensory Harvesting: Measured by the Nature Sensory Sensitivity Index (NSSI), a tool designed to quantify the objective capture of environmental stimuli.
2. Psychological Appraisal: Evaluated via the Perceived Restorativeness Scale (PRS).
3. Cognitive Function: Assessed through the Digit Span Task (Forward and Backward) to measure working memory and directed attention.
4. Affective States: Measured using the Profile of Mood States (POMS) to calculate Total Mood Disturbance (TMD) and self-esteem scales.
5. Physiological Response: Objective stress recovery was monitored via salivary cortisol levels and Heart Rate Variability (HRV), specifically the RMSSD (Root Mean Square of Successive Differences) to assess parasympathetic activation.

Statistical Analysis The study uses a serial mediation model to analyze how the environment intervention influences restorative outcomes through the sequential mediation of NSSI and PRS. Mixed-model ANOVAs are used to compare between-group differences across time points.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 30 years.
2. University students or individuals with equivalent educational background.
3. Normal or corrected-to-normal vision and hearing.
4. Willingness to comply with all study procedures and sign the informed consent form.

Exclusion Criteria:

1. Physical Health: History of cardiovascular disease, respiratory illness, or chronic pain that may affect Heart Rate Variability (HRV).
2. Mental Health: Diagnosis of clinical depression, anxiety disorders, or other psychiatric conditions.
3. Substance Use: Current smokers or individuals with a history of alcohol or drug abuse.
4. Medication: Recent use of any medications that affect the autonomic nervous system or endocrine function (e.g., steroids, beta-blockers, or hormonal medications) within the past month.
5. Cognitive/Physical Impairment: Any disability that prevents walking for 30 minutes or completing the Digit Span cognitive task.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Profile of Mood States - Total Mood Disturbance (ΔTMD) | From Baseline (Pre-test) to 30 minutes post-intervention (Post-test)
  The POMS TMD is a self-report scale consisting of 6 subscales: Tension, Depression, Anger, Fatigue, Confusion, and Vigor. Each item is rated on a 5-point scale (0 = Not at all to 4 = Extremely). The TMD score is calculated as: (Tension + Depression + Anger + Fatigue + Confusion) - Vigor. The final outcome (ΔTMD) is the difference between the post-intervention TMD score and the pre-intervention (baseline) TMD score [ΔTMD = TMD (Post) - TMD (Pre)]. TMD scores range from -120 to 120. A larger negative ΔTMD value indicates a greater reduction in negative emotions and more significant psychological restoration.

SECONDARY OUTCOMES:
Nature Relatedness (NR) | Baseline (T0, before intervention)
  This scale assesses the individual's levels of self-identification and connection with the natural world across three specific dimensions: NR-Self (e.g., "I feel that I am a part of nature"), NR-Experience (e.g., "I enjoy being outdoors, even in unpleasant weather"), and NR-Perspective (e.g., "Animals and plants should have rights similar to humans"). Items are rated on a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree). The Nature Relatedness (Final Score) is calculated as the average of all item scores. Total scores range from 6 to 30, where higher scores represent a stronger subjective connection and identification with nature.
Nature Sensory Sensitivity Index (NSSI) | Immediately after the 10-minute intervention (T1)
  The NSSI is a composite index designed to quantify objective and subjective sensory information harvesting across three sections:1. Section A: Free Recall: Participants have 2 minutes to list specific natural details perceived through sight, sound, smell, or touch. The score is the total number of valid natural items recalled.2. Section B: Sensory Recognition: A checklist of sensory items (e.g., fragrance of pine, rustling leaves) where participants tick items actually perceived. The score is the number of correct hits, excluding distractors (e.g., traffic noise).3. Section C: Aesthetic Immersion: A 3-item scale assessing immersion and "oneness" with the environment. Items are rated on a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree).The final NSSI score is a weighted composite of these three sections. The total score ranges from 0 to 100, higher scores indicate a greater volume, accuracy, and depth of sensory stimuli captured during the intervention.
Change in Perceived Restorativeness Scale (ΔPRS) | From Baseline (T0) to Immediately after the 10-minute intervention (T1)
  This scale assesses the participant's subjective perception of the environment's restorative qualities across four dimensions: Being Away, Fascination, Extent, and Compatibility. Each item is rated on a 5-point scale (1 = Not at all to 5 = Extremely). The final outcome (ΔPRS) is calculated as the difference between the post-intervention score and the pre-intervention baseline score [ΔPRS = PRS (Post) - PRS (Pre)]. The score for this change measure ranges from -4 to 4 (based on the average score difference). A positive ΔPRS indicates an increase in the perceived restorative quality of the environment.
Change in Total Digit Span Score (ΔDigit Span) | From Baseline (T0) to immediately after the 30-minute intervention (T2)
  This measure assesses the restoration of attention and working memory through two tasks: Digit Span Forward (Part A) and Digit Span Backward (Part B). For each task, participants are tested on span lengths from 3 to 9 digits, with two trials provided for each length. The Total Digit Span Score is the sum of the maximum spans or total successful trials from both tasks (A+B). The total score for this measure ranges from 0 to 18. The final outcome is the change score calculated as [ΔDigit Span = Digit Span (Post) - Digit Span (Pre)]. An increase in the score represents improved cognitive focus and restoration of directed attention.
Change in Self-Esteem (ΔSelf-Esteem) | From Baseline (T0) to immediately after the 30-minute intervention (T2)
  This scale measures the participant's state self-esteem and sense of self-worth based on their feelings "RIGHT NOW". It consists of 4 items assessing self-worth, positive qualities, attitude toward oneself, and self-satisfaction. Each item is rated on a 4-point scale (1=Strongly Disagree to 4=Agree). The total self-esteem score ranges from 4 to 16. The final outcome (ΔSelf-Esteem) is calculated as the difference between the post-intervention score and the pre-intervention baseline score [ΔSelf-Esteem = Self-Esteem (Post) - Self-Esteem (Pre)]. The score for this change measure ranges from -12 to 12. A positive ΔSelf-Esteem indicates an improvement in the individual's sense of self-worth following the intervention.

OTHER OUTCOMES:
Change in Heart Rate (ΔHR) | From Baseline (T0) to immediately after the 30-minute intervention (T2)
  This measure assesses the physiological stress recovery of participants by monitoring heart rate (measured in beats per minute, bpm). The final outcome is the change in heart rate calculated as [ΔHR = HR (Post) - HR (Pre)]. A decrease in heart rate from T0 to T2 indicates a transition toward parasympathetic nervous system dominance and successful physiological restoration.
Change in Salivary Cortisol (ΔCortisol) | From Baseline (T0) to immediately after the 30-minute intervention (T2)
  This measure assesses the biological stress response by measuring the concentration of cortisol in saliva, which reflects the activity of the Hypothalamic-Pituitary-Adrenal (HPA) axis. Saliva samples are collected using a swab and analyzed via enzyme-linked immunosorbent assay (ELISA). The concentration is typically measured in nmol/L or μg/dL. The final outcome is the change in cortisol levels calculated as [ΔCortisol = Cortisol (T2) - Cortisol (T0)]. A decrease in cortisol concentration indicates a reduction in physiological stress and a successful restorative effect of the environment.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, Study Director — Wuhan Technical University
Locations (1):
- Wuhan Technical University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to protect the privacy of the participants and ensure data security.